CLINICAL TRIAL: NCT03447275
Title: The Vitamin B Status in Type 2 Diabetes (VITA) Study
Acronym: VITA
Status: Completed | Type: Observational
Sponsor: Rima Obeid (Other)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry); Syneed Medidata GmbH (Industry)
Responsible Party: Sponsor-Investigator, Rima Obeid, Prof. Dr., Universität des Saarlandes
Organization: Universität des Saarlandes (Other)
Other Study IDs: EMR 200054-604
Record Dates: First submitted 2018-02-19; First posted 2018-02-27 (Actual); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Diabetes Mellitus, Type 2; Vitamin B 12 Deficiency; Vitamin B 6 Deficiency
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Vitamin B 12 Deficiency; Vitamin B 6 Deficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Controls: Apparently healthy subjects without type 2 diabetes
  Interventions: Other: Type 2 diabetes
- Patients with type 2 diabetes: type 2 Diabetes since 5 years or longer
  Interventions: Other: Type 2 diabetes

INTERVENTIONS:
Other: Type 2 diabetes — Test if patients with diabetes have different blood concentrations of vitamin biomarkers compared with control subjects and if vitamin levels in the patients will differ according to renal damage.

SUMMARY:
The objective of this study was to evaluate vitamin B deficiency (particularly vitamin B6 deficiency) in diabetic patients in Germany in relation to the presence or absence of proteinuria, and global vascular risk.

DETAILED DESCRIPTION:
This observational study recruited either control subjects or patients with type 2 diabetes for over 5 years and collected information on cardiovascular risk factors. Fasting blood samples and urine were collected and biomarkers of B-vitamins were measured and were related to renal function or to global cardiovascular risk. Global cardiovascular risk was calculated from established models that include Routine clinical and laboratory markers such as plasma lipids, smoking, hypertension, and BMI.

we measured the following markers: Glucose (fasting plasma glucose); HbA1C; serum creatinine; Glomerular filtration rate (GFR), urinary Albumin, C-reactive Protein, Soluble vascular cell adhesion molecule 1 (sVCAM-1), cystatin C, vitamin B1, vitamin B12, holotranscobalamin, methylmalonic acid, homocysteine, and different vitamin B6 forms.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent before any study-related activities
2. Ambulatory subject >18 years of age

   For patients with type 2 Diabetes:
3. Duration of diabetes ≥ 5 years
4. Glycated haemoglobin (HbA1C) <10%
5. Body mass index (BMI) 19-40 kg/m2

   For healthy controls:
6. No diabetes (normal fasting glucose levels measured by stick)

Exclusion Criteria:

1. End stage renal disease (creatinine clearance <10 mL/min)
2. Severe excess alcohol consumption (>50 units/week)
3. Severe co-morbidities
4. Renal and/or pancreatic transplant
5. Vitamin B1, B6 and/or B12 substitution (incl. multivitamin preparations)
6. Participation in an interventional study within 30 previous days;
7. Patient is female and pregnant or lactating
8. Patient is female in a childbearing age without adequate contraceptive precaution

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 122 patients with type 2 Diabetes and 52 control subjects were recruited (50% women in both groups).
Sampling Method: Probability Sample
Enrollment: 174 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
The difference in serum vitamin B12 levels between cases and controls | Baseline
  Compare mean levels of the controls with those in the patients
The difference in serum vitamin B1 between cases and controls | Baseline
  Compare mean levels of the controls with those in the patients
The difference in serum vitamin B6 concentrations between cases and controls | Baseline
  Compare mean levels of the controls with those in the patients

SECONDARY OUTCOMES:
The difference in serum vitamin B12 between patients with and those without albuminuria | Baseline
  Compare mean levels of diabetes patients with microalbuminuria and those without microalbuminuria
The difference in serum and urine vitamin B1 between patients with and those without albuminuria | Baseline
  Compare mean levels of diabetes patients with microalbuminuria and those without microalbuminuria
The difference in serum and urine vitamin B6 vitamers between patients with and those without albuminuria | Baseline
  Compare mean levels of diabetes patients with microalbuminuria and those without microalbuminuria
The difference in serum and urine vitamin B6 vitamers between patients with advanced global vascular risk versus those with a low vascular risk | Baseline
  Compare mean levels of diabetes patients with microalbuminuria and those without microalbuminuria

CONTACTS AND LOCATIONS:
Overall Officials: Wilfred A Nix, PhD, Principal Investigator — Department of Neurology, Medical University of Mainz, 55131 Mainz, Germany

IPD SHARING:
Plan to Share IPD: No
data will not be shared

REFERENCES:
- [Result] Nix WA, Zirwes R, Bangert V, Kaiser RP, Schilling M, Hostalek U, Obeid R. Vitamin B status in patients with type 2 diabetes mellitus with and without incipient nephropathy. Diabetes Res Clin Pract. 2015 Jan;107(1):157-65. doi: 10.1016/j.diabres.2014.09.058. Epub 2014 Oct 8. PMID 25458341
- See also: Journal Website — https://linkinghub.elsevier.com/retrieve/pii/S0168-8227(14)00458-6